CLINICAL TRIAL: NCT05962112
Title: Metabolic Implications of Day and Night-shift Working on NHS Healthcare Staff
Acronym: MIDNIGHT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 306915
Record Dates: First submitted 2023-05-23; First posted 2023-07-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-05

CONDITIONS: Shift-work Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Metabolic investigations after night-shifts — Metabolic investigations after night-shifts

SUMMARY:
The investigators will conduct an open label, experimental medicine study exploring the acute metabolic impact of night-shift compared to day-shift work in NHS healthcare workers. Employees who are scheduled to work both day and night shifts will be recruited and identical metabolic investigations will be performed in the same participant following at least 3 consecutive day and night-shifts respectively. These investigations will take place at the Clinical Research Unit (CRU) in Oxford Centre for Diabetes, Endocrinology and Metabolism (OCDEM) at Churchill Hospital. The order of post-day and post-night shift investigations will be randomly determined and there will be a 2-week minimum interval between both sets of investigations. Participants will complete a self-reported food diary before and during each set of shifts (both day and night) and will have wrist-watch actigraphy performed throughout the entire study period in order to measure sleep and activity parameters. All study visits and investigations will commence at the CRU at 8am and will include a 2-step hyperinsulinaemic euglycaemic clamp with stable isotope infusions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* National Health Service (NHS) worker with rotating night and day shift working patterns
* Age 18-75 years

Exclusion Criteria:

* A diagnosis of type 1 or type 2 diabetes
* Pregnancy
* A blood haemoglobin <120mg/dL
* History of alcohol use disorder or a greater than recommended alcohol intake (Recommendations > 21 units on average per week for men and > 14 units on average per week for women)
* Other conditions or co-morbidities that in the eyes of the investigators may affect data collection
* Any condition in the opinion of the investigator that might impact upon safety or validity of the results
* Primary sleep disorder
* Current glucocorticoid use
* Current melatonin use
* Patients with known non-alcoholic steatohepatitis or advanced hepatic fibrosis/cirrhosis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • NHS worker with rotating night and day shift working patterns
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in percentage incorporation of 2H2 palmitate from 2H2O into very low density lipoprotein triglyceride (VLDL-TG) after night shifts compared to day-shifts | Through study completion (average of 2 weeks)
  Incorporation of 2H2 palmitate from 2H2O into very low density lipoprotein triglyceride (VLDL-TG) represents a marker of hepatic de novo lipogenesis

SECONDARY OUTCOMES:
Change in hepatic and peripheral insulin sensitivity (measured by glucose metabolism during hyperinsulinaemic euglycaemic clamp procedure) after night shifts compared to day shifts | Through study completion (average of 2 weeks)
Mean daily sleep onset, wake time, midpoint of sleep, and sleep efficiency | Through study completion (average of 2 weeks)
  Measured by continuous actigraphy during night- compared to day-shifts night-shifts
Mean daily activity counts | Through study completion (average of 2 weeks)
  Measured by continuous wrist watch accelerometry during night- compared to day-shifts night-shifts

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No